CLINICAL TRIAL: NCT00997984
Title: A Phase 3, Double-blind, Randomized, Multicenter, Placebo-controlled, Dose Optimization Study Evaluating the Tolerability and Efficacy of AM and PM Once Daily Dosing With Extended-release Guanfacine Hydrochloride in Children Aged 6-12 With a Diagnosis of Attention-Deficit/Hyperactivity Disorder
Brief Title: Tolerability and Efficacy of AM and PM Once Daily Dosing With Extended-release Guanfacine Hydrochloride in Children 6-12 With Attention-Deficit/Hyperactivity Disorder (ADHD) (The ADHD Tempo Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD503-314
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Extended-release Guanfacine Hydrochloride (SPD503) AM (Experimental)
  Interventions: Drug: extended-release guanfacine hydrochloride (SPD503)
- placebo (Experimental)
  Interventions: Drug: placebo
- SPD503 PM (Experimental)
  Interventions: Drug: extended-release guanfacine hydrochloride

INTERVENTIONS:
Drug: extended-release guanfacine hydrochloride (SPD503) — dosed in AM
  Other Names: Intuniv
  Arms: Extended-release Guanfacine Hydrochloride (SPD503) AM
Drug: placebo — dosed in the AM or PM
  Arms: placebo
Drug: extended-release guanfacine hydrochloride — Dosed in the PM
  Other Names: Intuniv
  Arms: SPD503 PM

SUMMARY:
The primary purpose is to assess the efficacy of once daily dosing with optimized SPD503 (1, 2, 3 and 4mg/day), dosed either in the morning or evening, compared to placebo, in children with ADHD as measured by change from baseline score at endpoint on the ADHD-RS-IV.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years old
* ADHD diagnosis
* ADHD-RS-IV minimum score of 28
* CGI-S score > or = 4

Exclusion Criteria:

* Current, controlled or uncontrolled, comorbid psychiatric diagnosis
* Condition or illness which represent inappropriate risk to subject
* Known history or presence of structural cardiac abnormalities, serious heart rhythm abnormalities, syncope, cardiac conduction problems, exercise-related cardiac events, or clinically significant bradycardia; orthostatic hypotension or controlled or uncontrolled hypertension
* Use of prohibited medication that have CNS effects or affect cognitive performance
* History of alcohol or substance abuse within 6 months
* Current use of medication that affect BP or heart rate
* Significantly overweight
* Weight of less than 55 lbs
* Known allergy to SPD503
* Abnormal urine drug and alcohol screen

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2009-11-17 (Actual); Primary Completion 2010-10-09 (Actual); Study Completion 2010-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (46):
- United States (42):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Valley Clinical Research, Inc., El Centro, California
  - Peninsula Research Associates, Inc., Rolling Hills Estates, California
  - Psychiatric centers at San Diego, Feighner Research, San Diego, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Janus Centerfor Psychiatric Research, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northwest Clincial Research Group, Marietta, Georgia
  - Mountain West Clinical Trials, Boise, Idaho
  - University of Illinois Chicago, Chicago, Illinois
  - American Medical research, Inc., Oak Brook, Illinois
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Clinco, Terre Haute, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Marc Hertzman, M.D., P.C., Rockville, Maryland
  - Richester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Midwest research Group, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Children's Specialized Hospital, Toms River, New Jersey
  - Innovis Health, Fargo, North Dakota
  - IPS Research Company, Oklahoma City, Oklahoma
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Clinical Trials, Austin, Texas
  - Claghorn-Lesem research Clinic, Houston, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Western Clinical Investigations, Lubbock, Texas
  - Cerebral Research, LLC, San Antonio, Texas
  - Vermont Clinical Study Center, Burlington, Vermont
  - NeuroScience Inc, Herndon, Virginia
  - Alliance Research Group, LLC, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Canada (4):
  - BC Women;s Hospital and Health Centre, Vancouver, British Columbia
  - Toronto ADHD Clinic, Toronto, Ontario
  - ADHD Clinical/ The Kids Clinic, Whitby, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Newcorn JH, Stein MA, Childress AC, Youcha S, White C, Enright G, Rubin J. Randomized, double-blind trial of guanfacine extended release in children with attention-deficit/hyperactivity disorder: morning or evening administration. J Am Acad Child Adolesc Psychiatry. 2013 Sep;52(9):921-30. doi: 10.1016/j.jaac.2013.06.006. Epub 2013 Aug 1. PMID 23972694
- [Derived] Stein MA, Sikirica V, Weiss MD, Robertson B, Lyne A, Newcorn JH. Does Guanfacine Extended Release Impact Functional Impairment in Children with Attention-Deficit/Hyperactivity Disorder? Results from a Randomized Controlled Trial. CNS Drugs. 2015 Nov;29(11):953-62. doi: 10.1007/s40263-015-0291-6. PMID 26547425

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Dosed once daily in the morning (upon awakening) and once daily in the evening (7:00 PM)
- SPD503 AM: SPD503 dosed once daily at either 1, 2, 3 or 4 mg in the morning (upon awakening) and placebo dosed once daily in the PM (7:00 PM)
- SPD503 PM: Placebo dosed once daily in the AM (upon awakening) and SPD503 dosed once daily at either 1, 2, 3 or 4 mg in the PM (7:00 PM)
Period: Overall Study
Arm/Group | Placebo | SPD503 AM | SPD503 PM
Started | 113 | 113 | 114
Completed | 76 | 79 | 88
Not Completed | 37 | 34 | 26
Not completed — Adverse Event | 1 | 8 | 8
Not completed — Protocol Violation | 1 | 3 | 0
Not completed — Withdrawal by Subject | 6 | 9 | 5
Not completed — Lost to Follow-up | 8 | 5 | 4
Not completed — Lack of Efficacy | 20 | 6 | 3
Not completed — Met exclusion criteria | 1 | 0 | 0
Not completed — non-compliance | 0 | 2 | 3
Not completed — Wrong medication dispensed | 0 | 1 | 0
Not completed — Suicidal ideation | 0 | 0 | 1
Not completed — Work schedule | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SPD503 AM | SPD503 PM | Total
Number analyzed (Participants) | 112 | 107 | 114 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] — Based on the Full Analysis Set (FAS) defined as all subjects who had taken at least 1 dose of investigational product during the study. 340 subjects were randomized, but only 333 received at least 1 dose of investigational product.
  years | 8.9 (1.78) | 9.1 (1.77) | 9.3 (1.76) | 9.1 (1.77)
Age, Customized [Count of Participants; unit: Participants] — Based on the Full Analysis Set (FAS) defined as all subjects who had taken at least 1 dose of investigational product during the study. 340 subjects were randomized, but only 333 received at least 1 dose of investigational product.
  Participants
    6-12 years | 112 | 107 | 114 | 333
Sex: Female, Male [Count of Participants; unit: Participants] — Based on the Full Analysis Set (FAS) defined as all subjects who had taken at least 1 dose of investigational product during the study. 340 subjects were randomized, but only 333 received at least 1 dose of investigational product.
  Participants
    Female | 27 | 35 | 36 | 98
    Male | 85 | 72 | 78 | 235
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 110 | 104 | 110 | 324
  Canada | 2 | 3 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention-Deficit/Hyperactivity Disorder-Rating Scale-IV (ADHD-RS-IV) Total Score at Week 8 - Last Observation Carried Forward (LOCF)
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and up to 8 weeks
Population: Full Analysis Set (FAS) defined as all subjects who had taken at least 1 dose of investigational product during the study.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- All-Active: The combined results of the SPD503 AM and PM groups
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 110 | 104 | 111 | 215
Units on a scale | -10.6 (1.20) | -20.0 (1.23) | -20.4 (1.19) | -20.2 (0.86)
Statistical Analysis 1: Comparison: Placebo vs All-Active; Study designed to detect an effect size of 0.4 with 90% at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — A hierarchical testing structure was employed. First placebo vs all-active, then placebo vs am and lastly placebo vs pm. Testing was stopped when one comparison was not significant (p<0.05)
Statistical Analysis 2: Comparison: Placebo vs SPD503 AM; Study designed to detect an effect size of 0.4 with 90% at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs SPD503 PM; Study designed to detect an effect size of 0.4 with 90% at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Assessment of Clinical Global Impression-Severity of Illness (CGI-S) at Week 8 - LOCF
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: Baseline and up to 8 weeks
Population: FAS
Measure: Number; unit: Percent of Participants
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 110 | 104 | 112 | 216
Percent of Participants
  Normal, not at all ill | 4.5 | 11.5 | 16.1 | 13.9
  Borderline mentally ill | 8.2 | 20.2 | 20.5 | 20.4
  Mildly ill | 15.5 | 32.7 | 27.7 | 30.1
  Moderately ill | 34.5 | 22.1 | 22.3 | 22.2
  Markedly ill | 30.0 | 11.5 | 10.7 | 11.1
  Severely ill | 7.3 | 1.0 | 2.7 | 1.9
  Among the most extremely ill | 0.0 | 1.0 | 0.0 | 0.5
Statistical Analysis 1: Comparison: Placebo vs All-Active; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No formal adjustment for multiplicity was done
Statistical Analysis 2: Comparison: Placebo vs SPD503 AM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No formal adjustment for multiplicity was done
Statistical Analysis 3: Comparison: Placebo vs SPD503 PM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No formal adjustment for multiplicity was done

3. Secondary Outcome: Improvement on Clinical Global Impression-Improvement (CGI-I) Scale at Week 8 - LOCF
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement includes a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: up to 8 weeks
Population: FAS
Measure: Number; unit: Percent of Participants
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 110 | 104 | 112 | 216
Percent of Participants | 31.8 | 66.3 | 67.0 | 66.7
Statistical Analysis 1: Comparison: Placebo vs All-Active; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No formal adjustment for multiplicity was done
Statistical Analysis 2: Comparison: Placebo vs SPD503 AM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No formal adjustment for multiplicity was done
Statistical Analysis 3: Comparison: Placebo vs SPD503 PM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No formal adjustment for multiplicity was done

4. Secondary Outcome: Change From Baseline in Pediatric Daytime Sleepiness Scale (PDSS) Total Score at Week 8 - LOCF
Description: The Pediatric Daytime Sleepiness Scale (PDSS) is an 8 question questionnaire scored on a scale from 0 (never) to 4 (always). Total scores range from 0 to 32, with increasing score reflecting greater sleepiness.
Time Frame: Baseline and up to 8 weeks
Population: Safety Population defined as all subjects who had taken at least 1 dose of investigational product during the study.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 110 | 104 | 111 | 215
Units on a scale | -3.1 (0.53) | -2.7 (0.55) | -1.4 (0.53) | -2.0 (0.38)
Statistical Analysis 1: Comparison: Placebo vs All-Active; Test type: Superiority or Other; p = 0.099, ANCOVA — No formal adjustment for multiplicity was done
Statistical Analysis 2: Comparison: Placebo vs SPD503 AM; Test type: Superiority or Other; p = 0.596, ANCOVA — No formal adjustment for multiplicity was done
Statistical Analysis 3: Comparison: Placebo vs SPD503 PM; Test type: Superiority or Other; p = 0.023, ANCOVA — No formal adjustment for multiplicity was done

5. Secondary Outcome: Change From Baseline in Health Utilities Index-2/3 (HUI 2/3) Scores at Week 8 - LOCF
Description: HUI is used to describe health status and to obtain utility scores by collecting data using one or more questionnaires in formats selected to match the specific study design criteria. Scoring ranges from 0.00 (dead) to 1.00 (perfect health). Higher scores represent better health status.
Time Frame: Baseline and up to 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 99 | 97 | 100 | 197
Units on a scale | 0.043 (0.1159) | 0.056 (0.1166) | 0.063 (0.1100) | 0.060 (0.1131)

6. Secondary Outcome: Change From Baseline in Conner's Parent Rating Scale - Revised Short Version (CPRS-R:S) Score at Week 8 - LOCF
Description: The Conner's Parent rating Scale-revised short version (CPRS-R) consists of 27 questions graded on a scale from 0 (not true at all) to 3 (very much true) with a total score ranging from 0 to 81. Higher scores are indicative of increased ADHD. This scale allows parents to respond on the basis of the child's behavior and help assess ADHD and evaluate problem behavior.
Time Frame: Baseline and up to 8 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 86 | 87 | 91 | 178
Units on a scale | -10.4 (1.89) | -22.9 (1.88) | -21.2 (1.84) | -22.0 (1.31)
Statistical Analysis 1: Comparison: Placebo vs All-Active; Test type: Superiority or Other; p < 0.001, ANCOVA — No formal adjustment for multiplicity was done
Statistical Analysis 2: Comparison: Placebo vs SPD503 AM; Test type: Superiority or Other; p < 0.001, ANCOVA — No formal adjustment for multiplicity was done
Statistical Analysis 3: Comparison: Placebo vs SPD503 PM; Test type: Superiority or Other; p < 0.001, ANCOVA — No formal adjustment for multiplicity was done

7. Secondary Outcome: Change From Baseline in the Bedtime Resistance Subscale of Child's Sleep Habits Questionnaire (CSHQ) at Week 8 - LOCF
Description: The bedtime resistance subscale of CSHQ consists of 6 items scored on a scale from 1 (never/rarely) to 3 (Usually). A higher score reflects more disturbed sleep behavior.
Time Frame: Baseline and up to 8 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 109 | 103 | 111 | 214
Units on a scale | -0.7 (0.18) | -0.5 (0.18) | -1.0 (0.18) | -0.8 (0.13)
Statistical Analysis 1: Comparison: Placebo vs All-Active; Test type: Superiority or Other; p = 0.712, ANCOVA — No formal adjustment for multiplicity was done
Statistical Analysis 2: Comparison: Placebo vs SPD503 AM; Test type: Superiority or Other; p = 0.531, ANCOVA — No formal adjustment for multiplicity was done
Statistical Analysis 3: Comparison: Placebo vs SPD503 PM; Test type: Superiority or Other; p = 0.226, ANCOVA — No formal adjustment for multiplicity was done

8. Secondary Outcome: Post Sleep Questionnaire (PSQ) Quality of Sleep at Week 8 - LOCF
Description: Post Sleep Questionnaire (PSQ) overall rating of quality of sleep. There are 5 rating responses ranging from very poor to very good. No numbers are associated with the rating responses.
Time Frame: up to 8 weeks
Population: FAS
Measure: Number; unit: Percent of Participants
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 110 | 104 | 112 | 216
Percent of Participants
  Very poor | 2.7 | 1.0 | 0.0 | 0.5
  Poor | 6.4 | 5.8 | 7.1 | 6.5
  Average | 29.1 | 26.0 | 27.7 | 26.9
  Good | 35.5 | 42.3 | 50.9 | 46.8
  Very good | 26.4 | 25.0 | 14.3 | 19.4
Statistical Analysis 1: Comparison: Placebo vs All-Active; Test type: Superiority or Other; p = 0.859, Cochran-Mantel-Haenszel — No formal adjustment for multiplicity was done
Statistical Analysis 2: Comparison: Placebo vs SPD503 AM; Test type: Superiority or Other; p = 0.527, Cochran-Mantel-Haenszel — No formal adjustment for multiplicity was done
Statistical Analysis 3: Comparison: Placebo vs SPD503 PM; Test type: Superiority or Other; p = 0.739, Cochran-Mantel-Haenszel — No formal adjustment for multiplicity was done

9. Secondary Outcome: Change From Baseline in Mean Weiss Functional Impairment Rating Scale - Parent Report (WFIRS-P) Global Score at Week 8 - LOCF
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). Higher scores indicate greater functional impairment. Mean scores range from 0 to 3.
Time Frame: Baseline and up to 8 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 95 | 97 | 98 | 195
Units on a scale | -0.20 (0.038) | -0.35 (0.037) | -0.37 (0.037) | -0.36 (0.026)
Statistical Analysis 1: Comparison: Placebo vs All-Active; Test type: Superiority or Other; p < 0.001, ANCOVA — No formal adjustment for multiplicity was done
Statistical Analysis 2: Comparison: Placebo vs SPD503 AM; Test type: Superiority or Other; p = 0.004, ANCOVA — No formal adjustment for multiplicity was done
Statistical Analysis 3: Comparison: Placebo vs SPD503 PM; Test type: Superiority or Other; p = 0.001, ANCOVA — No formal adjustment for multiplicity was done

10. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week 8 - LOCF
Time Frame: Baseline and up to 8 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 110 | 104 | 112 | 216
mmHg
  Supine | -0.5 (9.39) | -1.6 (9.86) | -2.1 (10.26) | -1.9 (10.05)
  Standing | -1.4 (9.08) | -3.3 (11.23) | -2.7 (11.23) | -3.0 (11.20)
  Orthostatic | -0.9 (9.14) | -1.7 (9.89) | -0.6 (8.93) | -1.1 (9.40)

11. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 8 - LOCF
Time Frame: Baseline and up to 8 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 110 | 104 | 112 | 216
mmHg
  Supine | -0.3 (7.10) | -0.8 (7.98) | -2.1 (8.71) | -1.5 (8.37)
  Standing | 0.2 (7.74) | -2.2 (8.04) | -2.5 (9.91) | -2.4 (9.04)
  Orthostatic | 0.4 (6.31) | -1.4 (9.35) | -0.4 (8.94) | -0.9 (9.13)

12. Secondary Outcome: Change From Baseline in Pulse Rate at Week 8 - LOCF
Time Frame: Baseline and up to 8 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 110 | 104 | 112 | 216
beats per minute
  Supine | 1.0 (11.93) | -3.7 (12.35) | -3.8 (11.95) | -3.8 (12.12)
  Standing | 0.9 (12.02) | -1.9 (14.84) | -2.3 (11.41) | -2.1 (13.15)

13. Secondary Outcome: Change From Baseline in Oral Temperature at Week 8 - LOCF
Time Frame: Baseline and up to 8 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: º F
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 110 | 104 | 112 | 216
º F | 0.06 (0.779) | -0.12 (0.659) | -0.09 (0.758) | -0.10 (0.710)

14. Secondary Outcome: Change From Baseline in Height at Week 8 - LOCF
Time Frame: Baseline and up to 8 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 94 | 95 | 90 | 185
inches | 0.28 (0.412) | 0.39 (0.602) | 0.43 (0.459) | 0.41 (0.536)

15. Secondary Outcome: Change From Baseline in Weight at Week 8 - LOCF
Time Frame: Baseline and up to 8 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All-Active
Number analyzed (Participants) | 94 | 95 | 92 | 187
pounds | 2.15 (2.774) | 2.37 (2.684) | 2.64 (3.006) | 2.50 (2.843)

ADVERSE EVENTS:
Description: Safety Population defined as all subjects who had taken at least 1 dose of investigational product during the study.
Groups:
- All Active: The combined results of the SPD503 AM and PM groups
Arm/Group | Placebo | SPD503 AM | SPD503 PM | All Active
Serious Adverse Events (participants affected / at risk) | 0/112 | 1/107 | 2/114 | 3/221
Other Adverse Events (participants affected / at risk) | 64/112 | 85/107 | 95/114 | 180/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=112) | SPD503 AM (N=107) | SPD503 PM (N=114) | All Active (N=221)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2
Self-injurious ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=112) | SPD503 AM (N=107) | SPD503 PM (N=114) | All Active (N=221)
Somnolence (Nervous system disorders) | 14 | 50 | 48 | 98
Headache (Nervous system disorders) | 12 | 19 | 18 | 37
Sedation (Nervous system disorders) | 3 | 15 | 17 | 32
Abdomonal pain upper (Gastrointestinal disorders) | 8 | 7 | 20 | 27
Fatigue (General disorders) | 3 | 11 | 13 | 24
Irritability (General disorders) | 3 | 8 | 8 | 16
Nausea (Gastrointestinal disorders) | 1 | 6 | 6 | 12
Upper respiratory tract infection (Infections and infestations) | 11 | 8 | 4 | 12
Diarrhea (Gastrointestinal disorders) | 4 | 4 | 7 | 11
Dizziness (Nervous system disorders) | 3 | 6 | 5 | 11
Vomiting (Gastrointestinal disorders) | 2 | 7 | 4 | 11
Insomnia (Psychiatric disorders) | 4 | 6 | 3 | 9
Decreased appetite (Metabolism and nutrition disorders) | 3 | 6 | 3 | 9
Enuresis (Renal and urinary disorders) | 1 | 1 | 6 | 7
Increased appetite (Metabolism and nutrition disorders) | 6 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.